CLINICAL TRIAL: NCT01483261
Title: Is Trauma-Focused Cognitive Behavioral Therapy Effective in Reducing Post-traumatic Stress and Psychosocial Distress Among Sexually Exploited, War-affected Girls in the Democratic Republic of Congo.
Brief Title: An RCT of Trauma Focused-Cognitive Behavioral Therapy With Sexually Exploited, War-affected Girls in the DRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: World Vision (Other)
Responsible Party: Principal Investigator, Paul O'Callaghan, Doctoral Student in Educational, Child and Adolescent Psychology in Queen's University Belfast, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREC23-2011
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Post-traumatic Stress Symptoms; Psychosocial Distress
Keywords: Trauma-Focused Cognitive Behavior Therapy; Sexually Exploited Girls; Post-traumatic Stress Symptoms; Psychosocial Distress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma-Focused Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy
- Waiting List Control (No Intervention)

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — 15 sessions of manualised, culturally modified trauma-focused cognitive behavior therapy
  Arms: Trauma-Focused Cognitive Behavioral Therapy

SUMMARY:
To date, no RCT has examined the efficacy of Trauma-Focused Cognitive Behavioral Therapy with Sexually Exploited, War Affected Adolescent Girls in the Democratic Republic of Congo. This study seeks to fill this gap by designing, implementing and testing such an intervention using both an intervention and waiting list control group.

ELIGIBILITY:
Inclusion Criteria:

-Suicidal ideation (irrespective of score on any other measure)

Exclusion Criteria:

* psychosis
* mental retardation
* inability to understand Swahili
* one standard deviation below the mean on every measure

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in Post-traumatic Stress Symptoms as measured by the University of California Los Angelus Post Traumatic Stress Disorder -Reaction Index | baseline, post-intervention and 3-months

SECONDARY OUTCOMES:
Change in Psychosocial Distress as measured by the African Youth Psychosocial Assessment Instrument | baseline post-intervention and 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ciaran Shannon, BA, MA, DClin, Study Director — Chartered Clinical Psychologist (British Psychological Society)
Locations (1):
- World Vision Rebound Centre, Beni, South Kivu, Republic of the Congo

REFERENCES:
- [Derived] O'Callaghan P, McMullen J, Shannon C, Rafferty H, Black A. A randomized controlled trial of trauma-focused cognitive behavioral therapy for sexually exploited, war-affected Congolese girls. J Am Acad Child Adolesc Psychiatry. 2013 Apr;52(4):359-69. doi: 10.1016/j.jaac.2013.01.013. Epub 2013 Mar 6. PMID 23582867